CLINICAL TRIAL: NCT03794947
Title: Remote Ischaemic Conditioning for Fatigue After Stroke (RICFAST) - a Pilot, Double-blind, Randomised, Placebo Controlled Trial
Brief Title: Remote Ischaemic Conditioning for Fatigue After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH19508
Record Dates: First submitted 2018-11-29; First posted 2019-01-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Fatigue
Keywords: remote ischaemic conditioning
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischaemic Conditioning (Experimental): 4 cycles of 5 minutes of upper or lower (depending on tolerability) limb ischaemia followed by 5 minutes of reperfusion. This will be delivered using a manual shygnomanometer applied to the upper arm or leg and activated to go through 4 such cycles automatically. The blood pressure cuff in the active treatment arm will inflate to 200 mmHg (arm) and 220 mmHg (leg). RIC will be completed 3 times weekly for 4 weeks.
  Interventions: Procedure: Remote Ischaemic Conditioning
- Sham Intervention (Sham Comparator): 4 cycles of 5 minutes of upper or lower (depending on tolerability) limb ischaemia followed by 5 minutes of reperfusion. This will be delivered using a manual shygnomanometer applied to the upper arm or leg and activated to go through 4 such cycles automatically. The arm and leg blood pressure cuffs in the sham intervention will inflate to 20mmHg. Sham will be completed 3 times weekly for 4 weeks.
  Interventions: Procedure: Sham Intervention

INTERVENTIONS:
Procedure: Remote Ischaemic Conditioning — Induced ischaemia to a limb by inflating pressure cuffs around arms or legs to above systolic pressures (mmHg).
  Arms: Remote Ischaemic Conditioning
Procedure: Sham Intervention — The sham intervention will inflate pressure cuffs to much lower levels for the same number of cycles.
  Arms: Sham Intervention

SUMMARY:
This is a pilot randomised control trial to assess the safety, compliance, and acceptability of delivering a 6-week programme of remote ischaemic conditioning (RIC) to stroke patients suffering with fatigue, and study feasibility. A minimum of 34 patients who have suffered an ischeamic or haemorrhagic stroke and who suffer from fatigue, will be recruited and randomised to receive a 6-week programme of either RIC or a sham intervention.

DETAILED DESCRIPTION:
Up to 75% of stroke patients suffer from fatigue, the effect of which can be physical, cognitive or emotional, and presents a large barrier to progressing rehabilitation.

Remote ischaemic conditioning (RIC) is a procedure whereby ischaemia is induced to a limb for short periods of time by inflating pressure cuffs around arms or legs to above systolic pressures (mmHg). This procedure is performed for periods that avoid physical injury to the limbs, but induce neurohormonal, systemic or vascular changes in the body. Such changes often result in improved collateralisation of blood supply to various areas of the body, as well as improved efficiencies of cellular metabolism. This may enhance the physical abilities of patients undergoing rehabilitation after stroke, particularly when aiming to improve endurance and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged > 18 years) who have had an ischaemic or haemorrhagic stroke at least 6 weeks prior.
* Symptoms of debilitating fatigue for at least 4 weeks (fatigues severity score of 28 or more).

Exclusion Criteria:

* History or presence of significant peripheral vascular disease in the upper limbs.
* History or presence of complex neuropathic pains or peripheral neuropathy in the arms.
* Presence of lymphoedema in the arms.
* Presence of skin ulceration to the arms.
* Hospitalisation for cardiovascular or cerebrovascular disease within the last 4 weeks.
* Uncontrolled arrhythmia, hypertension, diabetes or angina.
* Third degree heart block or progressive heart failure.
* Acute aortic dissection, myocarditis, or pericarditis.
* Acute deep vein thrombosis, pulmonary embolism or pulmonary infection.
* Suspected or known dissecting aneurysm.
* Uncontrolled visual or vestibular disturbance.
* Known or suspected cause of fatigue e.g. obstructive sleep apnoea (Epworth > 15), depression (PHQ-9 > 14).
* Modified Rankin Score > 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Incidence of Treatment-Emergent Adverse Events. | 6 weeks
  Safety of a 6-week RIC intervention will be assessed by measuring the Number of Participants With Adverse Events That Are Related to Treatment.
% of RIC cycles completed | 6 weeks
  Compliance to RIC will be defined as achievement of 80% of intended RIC cycles. This will be assessed by a mobile compliance application.
Number of participants reporting RIC associated discomfort on a likert scale | 6 weeks
  Reported grade of discomfort associated with RIC will be measured on a likert scale of 0-5, 0 being no discomfort 5 being great discomfort. Acceptance of RIC will be defined as less than 1/3 of participants reporting moderate or greater discomfort (3-4 on scale) and will be supported by qualitative interviews and diary recordings.
number of participants recruited within the first 2 months | 1 year
  Study recruitment will be deemed feasible if four participants are recruited within the first 2 months.
Percentage of assessments completed | 1 year
  Study assessments will be deemed feasible if >80% of assessments are completed.

SECONDARY OUTCOMES:
Number of participants with abnormal changes from baseline in full blood count | 6 weeks
  Number of participants with changes to full blood count between baseline and after 6 week intervention period, leading to them lying outside the 'normal' range according to Sheffield Teaching Hospitals reference ranges. Any concerns or significant abnormalities will be referred to the principle investigator for appropriate action to ensure the safety of the participant.
number of participants with abnormal changes from baseline in urea and electrolyte (U&E) concentration | 6 weeks
  Number of participants with changes to U&E concentration between baseline and after 6 week intervention period, leading to them lying outside the 'normal' range according to Sheffield Teaching Hospitals reference ranges. Any concerns or significant abnormalities will be referred to the principle investigator for appropriate action to ensure the safety of the participant.
number of participants with abnormal changes from baseline in liver function | 6 weeks
  Number of participants with changes to liver function as measured by the liver function test (LFT) between baseline and after 6 week intervention period, leading to them lying outside the 'normal' range according to Sheffield Teaching Hospitals reference ranges. Any concerns or significant abnormalities will be referred to the principle investigator for appropriate action to ensure the safety of the participant.
Mean change from baseline in concentration of C-reactive protein (CRP) | 6 weeks
  The inflammatory marker (CRP) will be measured at baseline and after 6 week intervention period to assess if there has been a change in concentration between baseline and after the intervention.
Mean change from baseline in erythrocyte sedimentation rate (ESR) | 6 weeks
  ESR will be measured at baseline and after 6 week intervention period as a measure of inflammation.
Therapy Time in minutes | 6 weeks
  Measured at baseline and after 6 week intervention period.
Mean change from baseline in activity Energy Expenditure measure in kCal | 6 weeks
  Energy expenditure (kCal) will be measured using ACTiheart by CamnTech throughout the intervention period and changes from the baseline reviewed at the end of the 6 week intervention.
Mean change from baseline in minutes of activity per day measured by the Global Physical Activity Questionnaire (GPAQ) | 6 weeks
  The Global Physical Activity Questionnaire (GPAQ) measures physical activity levels from 3 domains: Activity at work, Travel to and from places, Recreational activities, as well as sedentary behaviour, in 16 questions, P1-P16. To analyse GPAQ data, metabolic equivalents (METs) are used to express the intensity of physical activities. MET is the ratio of a person's working relative to resting metabolic rate. Higher MET values indicate more intense activity. MET values are applied to time variables according to the intensity of the activity, 4 METS for time spent in moderate activities and 8 METS for vigorous activities. Mean/median time of physical activity on average per day is calculated by summing MET scores for all domains to calculate average activity per week, and dividing this score by 7 (p1t3+p4t6+p7t9+p10t12+p13t15)/7). The questionnaire will be completed at baseline and after 6 week intervention.
Mean change from baseline in distance walked as measured by the six minute walk test (6MWT) | 6 weeks
  The six minute walk test (6 MWT) is an exercise test that entails measurement of distance walked over a span of 6 minutes. Researcher will record the total distance walked, heart rate, blood pressure and Rating of Perceived Exertion (RPE). This will be done at baseline and after 6 week intervention period.
Mean change from baseline in peak oxygen consumption (VO2 max, ml/Kg/min) | 6 weeks
  At baseline and after 6 week intervention period.
Mean change from baseline in participant scores on the multidimensional fatigue inventory (MFI) | 6 weeks
  Measured with multidimensional fatigue inventory (MFI), a self report measure of fatigue. Participants indicate level of agreement with numerous statements associated with fatigue on a scale of 1-7, 1 being strongly disagree 7 being strongly agree. This is measured at baseline and after 6 week intervention period.
Mean change from baseline in participant scores on the modified rankin score (MRS) | 6 weeks
  Disability after stroke will be measured using modified rankin score (MRS), a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Symptoms are rated on a scale of 0 - 6, with 0 being 'no disability', rising in symptom severity to 6 being 'dead'. MRS will be taken at baseline and after 6 week intervention period.
Mean change from baseline in functional Independence as measured by the Barthel Index | 6 weeks
  Measured using Barthel Index (BI), an ordinal scale used to measure performance in 10 items (activities of daily living (ADL)). Items are rated on a scale from 0 - 15 in increments of 5, with 0 being least independent and 15 being most independent. Scores for all items are added up to give a total score out of 100, with higher scores equating to more independence. This is taken at baseline and after 6 week intervention period.
Mean change from baseline in depression as measured by participant scores on PHQ9 | 6 weeks
  Depression will be measured using Patient Health Questionnaire (PHQ9). The patient indicates how many times over the last two weeks have they been bothered by a series of 9 issues. The scale ranges from 0/not at all to 3/ nearly every day. Scores from each item are added to produce a final score out of 27, with scores 0-4 indicating no depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression and 20-27 severe depression. This is taken at baseline and after 6 week intervention period.
Mean change from baseline in anxiety as measured by participant scores on the GAD7 | 6 weeks
  Anxiety will be measured using the Generalised anxiety disorder assessment (GAD7). The patient indicates how many times over the last two weeks have they been bothered by a series of 7 issues. The scale ranges from 0/not at all to 3/ nearly every day. Scores from each item are added to produce a final score out of 21, Scores represent: 0-5 mild anxiety, 6-10 moderate anxiety, 11-15 moderately severe anxiety and 15-21 severe anxiety.This is taken at baseline and after 6 week intervention period.
Mean change from baseline in cognitive dysfunction as measured by participant scores on MOCA | 6 weeks
  Cognitive dysfunction will be measured using Montreal Cognitive Assessment (MOCA). This is a test with 8 domains, scores on each domain are added to produce a final score out of 30, with 26-30 equating to normal cognitive function. This will be completed at baseline and after 6 week intervention period.
Mean change from baseline in health related quality of life as measured by participant scores on EQ5D questionnaire. | 6 weeks
  Health Related Quality of Life will be measured by the EQ5D questionnaire at baseline and after 6 week intervention. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
Mean change from baseline in concentration of GLP-1 in blood sample | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, blood samples will be analysed for GLP-1 levels at baseline and after 6 week intervention.
Mean change from baseline in heat shock protein levels | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, blood samples will be analysed for heat shock protein levels at baseline and after 6 week intervention.
Changes from baseline in Cerebral Perfusion (ml/min) | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, changes in cerebral perfusion between baseline and after 6-week intervention period will be analysed.
Changes from baseline in levels of N-acetyl aspartate as measured by spectroscopy | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, changes in levels of tissue metabolite N-acetyl aspartate (that may indicate loss or damage to neuronal tissue) between baseline and after 6-week intervention period will be analysed.
Changes from baseline in levels of creatine as measured by spectroscopy | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, changes in levels of tissue metabolite creatine (that may indicate cell death through ischaemia) between baseline and after 6-week intervention period will be analysed.
Changes from baseline in levels of lactate as measured by spectroscopy | 6 weeks
  For a subset of patients who consent to having the MRI perfusion and spectroscopy studies as well as the blood analysis of biomarkers, changes in levels of tissue metabolite lactate between baseline and after 6-week intervention period will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ali, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT03794947/Prot_SAP_000.pdf